CLINICAL TRIAL: NCT02476526
Title: Safety of Low Dose Intravenous Contrast 64 Multi-Detector Computed Tomography Scanning in Patients With Chronic Kidney Disease
Brief Title: Safety of Low Dose IV Contrast CT Scanning in Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: General Electric (Industry)
Responsible Party: Principal Investigator, Bruce Barack, Section Chief, Thoracic Radiology, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Barack0001
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Chronic Kidney Disease; Pulmonary Embolism; Renal Artery Stenosis; Pulmonary Cancer
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pulmonary Embolism; Renal Artery Obstruction; Lung Neoplasms | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Volume Contrast (Experimental): Subjects in this arm will receive a single intravenous injection of low volume iso-osmolar non-ionic radio contrast medium, prior to undergoing 64-MDCT scanning. The use of low volume radio contrast medium constitutes the intervention. Both experimental and control groups receive a) acetylcysteine inhalation (Mucomyst) 1200 mg po BID x 48 hours starting the day prior to the CT scan; and b) isotonic Sodium Bicarbonate Solution 3ml/kg/hr iv for 1 hour prior to the CT scan and for 6 hours after the CT scan
  Interventions: Drug: Low Volume iso-osmolar non-ionic radio contrast medium; Drug: Acetylcysteine Inhalation; Drug: Sodium Bicarbonate Solution; Procedure: 64-MDCT Scanning
- Control (Sham Comparator): Subjects in this arm will undergo 64-MDCT scanning without Radio Contrast Medium (RCM). Both experimental and control groups receive a) acetylcysteine inhalation (Mucomyst) 1200 mg po BID x 48 hours starting the day prior to the CT scan; and b) isotonic Sodium Bicarbonate Solution 3ml/kg/hr iv for 1 hour prior to the CT scan and for 6 hours after the CT scan
  Interventions: Drug: Acetylcysteine Inhalation; Drug: Sodium Bicarbonate Solution; Procedure: 64-MDCT Scanning

INTERVENTIONS:
Drug: Low Volume iso-osmolar non-ionic radio contrast medium — Intravenous injection of low volume (30 cc) iso-osmolar non-ionic radio contrast medium as part of the 64-MDCT Scanning procedure (intervention group only)
  Other Names: Visipaque 320
  Arms: Low Volume Contrast
Drug: Acetylcysteine Inhalation — Mucomyst 1200 mg po BID x 48 hours starting the day prior to the CT scan (both experimental and control groups)
  Other Names: Mucomyst
Drug: Sodium Bicarbonate Solution — Isotonic Sodium Bicarbonate 3 ml/kg/hr iv for 1 hour prior to the CT scan and for 6 hours after the CT scan (both experimental and control groups)
  Other Names: Isotonic Sodium Bicarbonate
Procedure: 64-MDCT Scanning — Both experimental and control groups will undergo 64-MDCT scanning over the thoracic area
  Other Names: 64-Multi-Detector Computed Tomography Scanning

SUMMARY:
The purpose of this study is to show that the use of low volume iso-osmolar non-ionic radio contrast medium (30 cc) in a thoracic CT Scanning procedure in a selected group of patients with chronic kidney disease (CKD) will avoid contrast induced nephropathy (CIN) in comparison to a similar group of patients with CKD who receive no contrast medium..

DETAILED DESCRIPTION:
The use of radio contrast medium enhances the image quality of CT scans. However, contrast CT is avoided in patients with CKD for fear of contrast-induced nephropathy. The current standard of care for these patients is CT without contrast. Taking advantage of fast scanning capabilities of modern CT scanners (64-Multi-Detector CT), the current investigators have developed a method to use low volume iso-osmolar non-ionic radio contrast medium (30 cc) which can be used in a selected group of adult patients with mild to moderate stable CKD (eGFR 16-60 ml/min/m^2 for at least 12 months), who require thoracic CT imaging for diagnostic purposes. Up to 100 patients who meet the inclusion/exclusion criteria will be randomized to standard care (no-contrast, 50 controls) or low volume contrast CT (50 intervention group). The peak increase of serum creatinine levels within 72 hours after the CT procedure will be measured as an outcome variable for comparison between the two groups, as well as a safety monitoring variable in the intervention group (25% increase is the upper threshold).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented stable Chronic Kidney Disease (CKD) defined as a stable eGFR 16-60 ml/min/m^2 for ≥ 12 months; and
* Referred to CT scanning procedure to evaluate pulmonary embolism, pulmonary malignancy, acute aortic syndromes, or renal artery stenosis.

Exclusion Criteria:

* CKD Stages 1, 2 and 5
* Stage 3-4 congestive heart failure (CHF)
* Irregular supraventricular tachycardia
* Allergic to iodinated Radio Contrast Medium (RCM)
* Allergic to Mucomyst
* Pregnancy
* Evidence of acute renal failure (ARF)
* Serum bicarbonate either less than 20 meq/L or greater than 35 meq/L
* Hydration with a bicarbonate solution is contraindicated or considered unsafe by the subject's caring physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Peak Serum Creatinine Level | Up to 72 hours after intervention
  The peak serum creatinine increase over baseline within 72 hours after intervention is the outcome variable. This variable is used for comparison between two groups, as well as for safety monitoring in the intervention group (25% increase is the upper threshold)

CONTACTS AND LOCATIONS:
Overall Officials: Dean T Yamaguchi, MD, PhD, Study Director — VA Greater Los Angeles Healthcare System
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Results will be published after completion of study.

REFERENCES:
- [Background] Levey AS, Coresh J, Balk E, Kausz AT, Levin A, Steffes MW, Hogg RJ, Perrone RD, Lau J, Eknoyan G; National Kidney Foundation. National Kidney Foundation practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Ann Intern Med. 2003 Jul 15;139(2):137-47. doi: 10.7326/0003-4819-139-2-200307150-00013. PMID 12859163